CLINICAL TRIAL: NCT06944990
Title: Meta Self-efficacy Intervention to Improve Work Self-efficacy and Occupational Well-being in Young Employees: Internet Intervention Co-creation and a Randomized Controlled Trial
Brief Title: Meta Self-efficacy Internet Intervention to Improve Work Self-efficacy and Occupational Well-being in Young Employees
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Principal Investigator, Jan Maciejewski, Principal Investigator, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSE intervention
Record Dates: First submitted 2025-04-11; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Self Efficacy; Occupational Stress; Well-Being, Psychological; Work Related Stress
Keywords: meta self-efficacy; self-efficacy; job affective well-being; sustainable employability; work stress; work self-efficacy
MeSH Terms: conditions — Occupational Stress; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Masking Description: Group allocation will not be disclosed to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meta self-efficacy internet intervention (Experimental): The meta self-efficacy intervention is a three-week program comprised of activities designed to enhance meta self-efficacy (the ability to leverage self-efficacy sources). The intervention is contextualized to young employees.
  Interventions: Behavioral: Meta self-efficacy internet intervention
- Placebo (Placebo Comparator): The placebo condition contains educational material delivered with the same modality as in the experimental condition.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Meta self-efficacy internet intervention — The meta self-efficacy intervention is a three-week program comprised of activities designed to enhance meta self-efficacy (the ability to leverage self-efficacy sources). The intervention is contextualized to young employees.
  Arms: Meta self-efficacy internet intervention
Behavioral: Placebo — The placebo condition contains educational material delivered with the same modality as in the experimental condition.
  Arms: Placebo

SUMMARY:
This randomized controlled trial aims to test whether enhancing meta self-efficacy through a self-guided internet intervention improves young employees' work self-efficacy and occupational well-being. The trial will evaluate primary (work self-efficacy) and secondary (three dimensions of occupational well-being) outcomes. It is hypothesized that boosting meta self-efficacy will lead to improvements in outcomes, with effects assessed immediately after the intervention, and at 3- and 6-month follow-ups.

DETAILED DESCRIPTION:
This study investigates the efficacy of a self-guided internet intervention designed to enhance meta self-efficacy in young employees. Meta self-efficacy is a psychological resource that encompasses the ability to leverage self-efficacy sources (mastery experiences, vicarious experiences, persuasion, and affective & physiological states) to boost context-specific self-efficacy. In this two-arm randomized controlled trial, participants (young employees) will be randomly assigned to an experimental group, which will receive internet intervention with activities aimed at enhancing meta self-efficacy, or to a placebo control group, which will receive educational content. Primary and secondary outcomes (including work self-efficacy, job stress, job affective well-being, and work capabilities), as well as the manipulation check (meta self-efficacy), will be assessed immediately after the intervention and at 3- and 6-month follow-ups. The trial aims to evaluate the effect of enhancing meta self-efficacy and explore the impact of factors such as adherence and engagement on the intervention's efficacy.

ELIGIBILITY:
Inclusion Criteria:

* must be between 18 and 30 years old
* must be empolyed (working at least 20 h / week, for at least the prior two months, regardless of the type of contract)

Exclusion Criteria:

* none

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Work Self-Efficacy | Posttest (after 3 weeks), 3-months follow-up, 6-months follow-up
  Work Self-Efficacy will be measured with the Work Self-Efficacy scale (WSES). The questionnaire consists of 26 items. The responses range from 1 (not at all) to 7 (completely).

SECONDARY OUTCOMES:
Job Affective Well-Being | Posttest (after 3 weeks), 3-months follow-up, 6-months follow-up
  Job Affective Well-Being will be measured with the Job Affective Well-Being Scale (JAWS). The questionaire consists of 12 items. The responses rage from 1 (never) to 5 (very often).
Job Stress | Posttest (after 3 weeks), 3-months follow-up, 6-months follow-up
  Job Stress will be measured with the Perceived Stress Scale (PSS). The scale consists of 4 items rated on a scale ranging from 0 (never) to 4 (very often). It will be applied to measure job stress. The questionnaire's instructions have been modified to align with the occupational context.
Work Capabilities | Posttest (after 3 weeks), 3-months follow-up, 6-months follow-up
  Work capabilities will be measured with the Capability Set for Work Questionaire (CSWQ). The questionaire consists of 7 capabilities, for each there are three aspects to evaluate. The responses range from 1 (strongly disagree) to 5 (strongly agree).

OTHER OUTCOMES:
Meta self-efficacy. | Posttest (after 3 weeks), 3-months follow-up, 6-months follow-up
  Meta self-efficacy will be measured with the meta self-efficacy scale (MSES). The questionnaire consists of 13 items. The responses range from 0 (cannot do at all) to 10 (certain can do). Higher score indicates higher level of meta self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Maciejewski, Principal Investigator — SWPS University
Locations (1):
- SWPS University of Social Sciences and Humanities, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Smoktunowicz E, Lesnierowska M, Carlbring P, Andersson G, Cieslak R. Resource-Based Internet Intervention (Med-Stress) to Improve Well-Being Among Medical Professionals: Randomized Controlled Trial. J Med Internet Res. 2021 Jan 11;23(1):e21445. doi: 10.2196/21445. PMID 33427674
- [Derived] Maciejewski J, Cieslak R, Carlbring P, Smoktunowicz E. Meta Self-Efficacy Internet Intervention to Support Occupational Health in Young Employees: Protocol for Co-Creation and a Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 23;14:e85082. doi: 10.2196/85082. PMID 41432307